CLINICAL TRIAL: NCT05470114
Title: A Randomized, Double-blinded, Active Comparator-controlled, 16-week, Single-site, Exploratory, Mechanistic Trial to Assess the Effect of LEO 138559 on the Molecular Signature and Safety in Adults With Moderate to Severe Atopic Dermatitis.
Brief Title: A Multi-omics Disease Signature Trial in Adult Patients With Moderate to Severe AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0145-2274; 2021-006211-28 (EudraCT Number)
Record Dates: First submitted 2022-05-19; First posted 2022-07-22 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEO 138559 (Experimental): Participants received injections of LEO 138559 from Week 0 (baseline) to Week 16 (end of treatment).
  Interventions: Drug: LEO 138559
- Dupixent® (Active Comparator): Participants received injections of Dupixent® from Week 0 (baseline) to Week 16 (end of treatment).
  Interventions: Drug: Dupixent®

INTERVENTIONS:
Drug: LEO 138559 — LEO 138559 is an antibody given by subcutaneous injection.
  Arms: LEO 138559
Drug: Dupixent® — Dupixent® is an antibody given by subcutaneous injection.
  Arms: Dupixent®

SUMMARY:
This clinical trial will investigate the effectiveness and safety of a new active ingredient (LEO 138559) in the treatment of moderate to severe atopic dermatitis (AD). It is given by subcutaneous injection. Some people in the trial will instead receive Dupixent® which is an approved treatment for moderate to severe AD. Dupixent® is also given by subcutaneous injection.

The main aim of this clinical trial is to investigate which changes in biomarkers in the skin are caused by LEO 138559 and Dupixent®.

The trial includes a screening phase of up to 4 weeks, followed by a treatment period of 16 weeks, and a safety follow-up period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD [as defined by the American Academy of Dermatology (AAD) Consensus Criteria] that has been present for ≥1 year prior to screening.
* Subjects who have a recent history (within 6 months before screening) of inadequate response to treatment with topical medication, or for whom topical treatments are otherwise medically inadvisable.
* EASI score ≥12 at screening and ≥16 at baseline.
* vIGA-AD score ≥3 at screening and baseline.
* Body surface area (BSA) of AD involvement ≥10% at screening and baseline.
* Worst Daily Pruritus NRS (weekly average) of ≥3 points at baseline.

Exclusion Criteria:

* Treatment with systemic immunosuppressive/immunomodulating medication (excluding systemic antihistamines if taken at stable dose already before baseline), e.g., JAK inhibitors, immunoglobulin/blood products, or phototherapy within 4 weeks or 5 half-lives prior to baseline, whichever is longer.
* Treatment with systemic corticosteroids within 4 weeks prior to baseline (NOTE: Inhaled or intranasal steroids equivalent to doses including and up to 500 µg beclometasone (or equivalent) daily is allowed).
* Treatment with biologics within 5 half-lives (if known) or 16 weeks prior to baseline, whichever is longer.
* Treatment with TCS, TCI, or topical PDE-4 inhibitor within 1 week prior to baseline (NOTE: Patient may be rescreened (one time) if failed for this criterion.
* Intake of nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 week prior to baseline. Intake of paracetamol will be allowed.
* Treatment with a live (attenuated) vaccine within 12 weeks prior to baseline.
* Clinically significant active chronic or acute infection requiring systemic treatment within 4 weeks prior to baseline that may compromise the safety of the subject.
* Clinically significant abnormalities detected on vital signs or ECG (apart from 1st degree atrioventricular (AV) block that is allowed).
* Serious heart conditions, chronic lung diseases.
* Acute asthma, acute bronchospasm, moderate to severe asthma.
* Skin infection within 1 week prior to the baseline visit.
* Presence of hepatitis B or C infection at screening.
* Active inflammatory bowel disease (IBD) or history of IBD, anaphylaxis, immune complex disease, pancreatic disease, zoster infections, viral skin infections (including eczema herpeticum) or known or suspected history of immunosuppressive disorder.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Subject has a positive test for tuberculosis at screening.
* Subject is pregnant or lactating.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Investigational Site, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LEO 138559: Participants will receive injections of LEO 138559 from Week 0 (baseline) to Week 16 (end of treatment).
  LEO 138559: LEO 138559 is an antibody given by subcutaneous injection.
- Dupixent®: Participants will receive injections of Dupixent® from Week 0 (baseline) to Week 16 (end of treatment).
  Dupixent®: Dupixent® is an antibody given by subcutaneous injection.
Period: Overall Study
Arm/Group | LEO 138559 | Dupixent®
Started | 9 | 4
Completed | 7 | 4
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 138559 | Dupixent® | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (11.3) | 26.0 (5.9) | 30.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 9 | 4 | 13
Baseline height (cm) [Mean (Standard Deviation); unit: cm] | 176.1 (11.1) | 171.0 (4.7) | 174.5 (9.7)
Baseline weight (kg) [Mean (Standard Deviation); unit: kg] | 82.49 (13.61) | 71.75 (9.98) | 79.18 (13.23)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gene Expression Typically Associated With Atopic Dermatitis in Lesional Skin Biopsies From Baseline to Week 4
Description: Lesional skin biopsies will be evaluated by single cell RNA sequencing to evaluate global gene expression
Time Frame: From baseline to week 4
Population: The analysis population consists of individuals with AD, and the gene expression analysis is based on lesional skin biopsies obtained from these individuals at baseline and week 4. The gene expression values used in the analysis are averaged expression values for each identity class. These values were calculated using the AverageExpression function on the basis of normalized data from the respective Seurat object.
  In LEO 138559 Arm group, 1 participant screened but not included in the analysis.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | LEO 138559 | Dupixent®
Number analyzed (Participants) | 8 | 4
fold change
  Keratinocytes S100A7 | 0.212 (7.692) | 0.043 (8.899)
  Keratinocytes S100A8 | 0.155 (6.308) | 0.048 (5.367)
  Keratinocytes S100A9 | 0.149 (5.52) | 0.02 (13.99)
  Keratinocytes KRT6A | 0.164 (4.08) | 0.088 (1.459)
  Keratinocytes KRT16 | 0.246 (2.75) | 0.094 (1.731)
  Keratinocytes KRT1 | 1.355 (1.748) | 0.851 (5.008)

2. Secondary Outcome: Number of Treatment-emergent Adverse Events From Baseline to Week 16 Per Subject
Time Frame: Between baseline and week 16
Measure: Number; unit: Events
Arm/Group | LEO 138559 | Dupixent®
Number analyzed (Participants) | 9 | 4
Events | 17 | 8

ADVERSE EVENTS:
Time Frame: Baseline to 16 week
Arm/Group | LEO 138559 | Dupixent®
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 8/9 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 138559 (N=9) | Dupixent® (N=4)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Malassezia infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT05470114/Prot_SAP_000.pdf